CLINICAL TRIAL: NCT00924469
Title: A Phase 2 Open-Label, Randomized, Multi-center Study of Neoadjuvant Abiraterone Acetate (CB7630) Plus Leuprolide Acetate and Prednisone Versus Leuprolide Acetate Alone in Men With Localized High Risk Prostate Cancer
Brief Title: A Phase 2 Study to Evaluate Safety and Efficacy of Abiraterone Acetate in Male Participants With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016936; COU-AA-201 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Abiraterone acetate; Leuprolide acetate; Prednisone; CB7630; Testosterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; Leuprolide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abiraterone plus leuprolide plus prednisone (Experimental): Abiraterone acetate tablets will be administered orally at a total dose of 1000 milligram (mg) per day up to Week 24. Leuprolide acetate will be administered at a dose of 22.5 mg (dose adjusted as per Investigator's discretion) as intramuscular injection (injection of a substance into a muscle) once every 12 weeks up to Week 24. Prednisone tablets will be administered orally as 5 mg once daily for 24 weeks.
  Interventions: Drug: Abiraterone; Drug: Leuprolide; Drug: Prednisone
- Leuprolide then abiraterone plus leuprolide plus prednisone (Active Comparator): Leuprolide acetate will be administered at a dose of 22.5 mg as intramuscular injection once every 12 weeks up to Week 24. From Week 13 to 24, abiraterone acetate tablets will be administered orally at a total dose of 1000 mg per day with prednisone tablets administered orally as 5 mg once daily.
  Interventions: Drug: Abiraterone; Drug: Leuprolide; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone — Abiraterone acetate tablets will be administered orally at a total dose of 1000 milligram (mg) per day at least 1 hour before a meal or 2 hours after a meal for 24 weeks in Group 1 and from Week 13 to Week 24 for Group 2.
  Other Names: CB7630
Drug: Leuprolide — Leuprolide acetate will be administered at a dose of 22.5 mg (dose adjusted as per Investigator's discretion) as intramuscular injection (injection of a substance into a muscle) once every 12 weeks in Group 1 and Group 2.
Drug: Prednisone — Prednisone tablets will be administered orally as 5 mg once daily for 24 weeks in Group 1 and from Week 13 to Week 24 for Group 2.

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of abiraterone acetate plus leuprolide acetate and prednisone, versus leuprolide acetate alone in male participants with prostate cancer (a disease in which cells in the prostate gland become abnormal and start to grow uncontrollably, forming tumors) who are suitable candidates for prostatectomy (surgery to remove all or part of the prostate gland).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study drug is assigned by chance), and multi-center (conducted in more than one center) study of abiraterone in male participants with prostate cancer. The duration of study will be approximately 24-32 weeks per participant. The study consists of 4 parts: Screening (that is, 30 days before study commences on Day 1); Treatment (abiraterone acetate 1000 milligram per day or leuprolide acetate as 22.5 milligram intramuscular injection [injection of a substance into a muscle] or prednisone 5 mg once daily); Prostatectomy (Week 24); and Follow-up ( 4-8 weeks after prostatectomy). Participants will receive either abiraterone, leuprolide and prednisone for 24 weeks (that is, Group 1) or leuprolide once every 12 weeks up to Week 24 then abiraterone and prednisone from Week 13 to 24 (that is, Group 2). All the eligible participants will be randomly assigned to 1 of the 2 treatment groups. Efficacy will be evaluated primarily through the concentrations of testosterone and dihydrotestosterone from prostate tissues at Week 12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* At least three core biopsies positive for prostate cancer (a minimum of 6 core biopsies must be obtained at baseline). A prostate biopsy within 6 months from Screening is allowed for entry requirements
* At least one of the following features: prostate specific antigen (PSA) greater than (>) 10 nanogram per milliliter (ng/ml); PSA velocity >2 ng/ml per /year (defined as a rise in PSA of >2 ng/ml in the preceding 12 month period); Gleason score greater than or equal to (>=) 7 (4+3); Gleason score 6 if either PSA >=10 ng/ml or PSA velocity >=2 ng/ml/year
* Serum testosterone >200 nanogram/deciliter
* Participant and urologist must agree that participant is suitable for prostatectomy

Exclusion Criteria:

* Serious or uncontrolled co-existent, non-malignant disease, including active and uncontrolled infection
* Abnormal liver function consisting of any of the following: serum bilirubin >= 1.5 * upper limit of normal (ULN); aspartate aminotransferase or alanine aminotransferase >=2.5 * ULN
* Uncontrolled hypertension within the Screening period (systolic blood pressure >= 160 millimeter of mercury [mmHg] or diastolic BP >= 95 mmHg)
* Requirement for corticosteroids greater than the equivalent of 5 milligram of prednisone daily
* Participants with active or symptomatic viral hepatitis or chronic liver disease or clinically significant heart disease or as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50 percent at Baseline or history of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug or history of pituitary or adrenal dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Boston, Massachusetts
  - Houston, Texas
  - Seattle, Washington
  - Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Plus Leuprolide Plus Prednisone: Abiraterone acetate tablets were administered orally at a total dose of 1000 milligram (mg) per day up to Week 24. Leuprolide acetate was administered at a dose of 22.5 mg (dose adjusted as per Investigator's discretion) as intramuscular injection (injection of a substance into a muscle) once every 12 weeks up to Week 24. Prednisone was administered orally as 5 mg tablets once daily for 24 weeks.
- Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone: Leuprolide acetate was administered at a dose of 22.5 mg as intramuscular injection once every 12 weeks up to Week 24. From Week 13 to 24, abiraterone acetate tablets were administered orally at a total dose of 1000 mg per day with prednisone administered orally as 5 mg tablets once daily.
Period: Overall Study
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Started | 30 | 28
Completed | 28 | 26
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone | Total
Number analyzed (Participants) | 30 | 28 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 61.0 (6.67) | 56.9 (5.30) | 59.0 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Testosterone Concentration in Prostate Tissue
Description: Testosterone is a potent androgen (a hormone that promotes the development and maintenance of male characteristics) and major product secreted by cells in the testis and produced in the adrenal glands and by prostate cancers. Abiraterone acetate affects sources of testosterone in the body (ie, adrendal gland and prostate tumor). Testosterone concentration was measured in prostate tissues after exposure to study treatments at Week 12.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all the participants who were randomly assigned to the study treatment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Picogram per milligram (pg/mg)
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 28 | 27
Picogram per milligram (pg/mg) | 0.089 (0.0637) | 0.228 (0.3788)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for testosterone concentration at Week 12; Test type: Superiority or Other; p = 0.0216, ANOVA — Test for no difference of natural log transformed values between treatments was calculated using two-way analysis of variance (ANOVA) adjusting for Baseline risk factor; Adjusted mean ratio = 0.61, 90% CI [0.429 to 0.865]

2. Secondary Outcome: Testosterone and Dihydrotestosterone (DHT) Concentration in Prostate Tissue
Description: Testosterone is a potent androgen (a hormone that promotes the development and maintenance of male characteristics) and major product secreted by cells in the testis and produced in the adrenal glands and by prostate cancers. Dihydrotestosterone (DHT) is a potent androgenic metabolite of testosterone. Testosterone and DHT concentration was measured in prostate tissues after exposure to study treatments at Week 24.
Time Frame: Week 24
Population: ITT population included all the participants who were randomly assigned to the study treatment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Picogram per milligram (pg/mg)
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 28 | 26
Picogram per milligram (pg/mg)
  Testosterone | 0.216 (0.6707) | 0.062 (0.0340)
  DHT | 1.340 (3.5099) | 2.456 (6.3901)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for testosterone concentration at Week 24; Test type: Superiority or Other; p = 0.1423, ANOVA — Test for no difference of natural log transformed values between treatments was calculated using two-way ANOVA adjusting for Baseline risk factor; Adjusted mean ratio = 1.43, 90% CI [0.956 to 2.145]
Statistical Analysis 2: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 2 for DHT concentration at Week 24; Test type: Superiority or Other; p = 0.6639, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 0.82, 90% CI [0.386 to 1.746]

3. Secondary Outcome: Androstenedione and Dehydroepiandrosterone (DHEA) Concentrations in Prostate Tissue
Description: Androstenedione is a steroid (a group of polycyclic compounds closely related biochemically to terpenes, for example, cholesterol, numerous hormones), that is produced in the testis, ovary and the adrenal cortex, and depending on the tissue type, androstenedione can serve as a precursor to testosterone, estrone and estradiol. The DHEA is a major steroid produced by the adrenal cortex. It is also produced in small quantities in the testis and the ovary. Androstenedione and DHEA concentration was measured in prostate tissues at Week 12 and 24.
Time Frame: Week 12 and 24
Population: ITT population included all the participants who were randomly assigned to the study treatment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure and "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Picogram per milligram (pg/mg)
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 28 | 27
Picogram per milligram (pg/mg)
  Androstenedione: Week 12 (n=28,27) | 0.082 (0.0525) | 0.277 (0.1729)
  Androstenedione: Week 24 (n=28,26) | 0.090 (0.0879) | 0.070 (0.0403)
  DHEA: Week 12 (n=28,27) | 1.994 (5.0266) | 29.241 (26.9800)
  DHEA: Week 24 (n=28,26) | 3.138 (8.6692) | 2.170 (3.7095)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for androstenedione concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 0.32, 90% CI [0.239 to 0.418]
Statistical Analysis 2: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 2 for androstenedione concentration at Week 24; Test type: Superiority or Other; p = 0.5061, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 1.13, 90% CI [0.828 to 1.554]
Statistical Analysis 3: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 3 for DHEA concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 0.03, 90% CI [0.017 to 0.050]
Statistical Analysis 4: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 4 for DHEA concentration at Week 24; Test type: Superiority or Other; p = 0.5767, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 0.79, 90% CI [0.398 to 1.581]

4. Secondary Outcome: Serum Levels of Androgens
Description: Serum concentrations of testosterone, DHT, androsterone, DHEA, DHEA-Sulfate, DHEA-Glucuronide and delta-4-androstenedione were measured at Weeks 12 and 24.
Time Frame: Week 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Nanogram per deciliter (ng/dL)
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 29 | 28
Nanogram per deciliter (ng/dL)
  Testosterone: Week 12 (n=28,28) | 1.049 (1.0374) | 10.014 (12.5981)
  Testosterone: Week 24 (n=25,25) | 0.648 (0.4975) | 3.122 (12.6460)
  DHT: Week 12 (n=28,28) | 6.143 (8.9868) | 5.797 (5.9816)
  DHT: Week 24 (n=26,26) | 5.932 (9.1599) | 6.730 (15.7929)
  Androsterone: Week 12 (n=28,28) | 0.619 (0.4473) | 3.100 (5.8891)
  Androsterone: Week 24 (26,26) | 1.752 (6.3226) | 0.500 (0.0000)
  DHEA: Week 12 (n=28,28) | 10.684 (27.2814) | 180.307 (133.6277)
  DHEA: Week 24 (n=26,26) | 20.922 (64.2594) | 7.617 (14.5386)
  DHEA-Glucuronide: Week 12 (n=29,28) | 69.724 (184.2399) | 583.036 (879.7514)
  DHEA-Glucuronide: Week 24 (n=27,27) | 51.675 (148.9412) | 51.759 (95.0666)
  DHEA-Sulfate: Week 12 (n=28,28) | 7156.270 (22406.7048) | 133338.875 (108819.6403)
  DHEA-Sulfate: Week 24 (n=26,26) | 9047.406 (27844.7883) | 9207.345 (30897.5488)
  Delta-4-Androstenedione:Week 12(n=28,28) | 3.315 (3.3858) | 33.330 (26.8110)
  Delta-4-Androstenedione:Week 24(n=26,26) | 5.192 (10.8654) | 2.831 (1.1596)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for serum testosterone concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test for no difference of natural log transformed values between treatments was calculated using analysis of covariance (ANCOVA) adjusting for Baseline risk factor and Baseline androgen; Adjusted mean ratio = 0.14, 90% CI [0.097 to 0.207]
Statistical Analysis 2: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 2 for serum testosterone concentration at Week 24; Test type: Superiority or Other; p = 0.4364, ANCOVA — Test for no difference of natural log transformed values between treatments was calculated using ANCOVA adjusting for Baseline risk factor and Baseline androgen; Adjusted mean ratio = 0.84, 90% CI [0.571 to 1.225]
Statistical Analysis 3: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 3 for serum DHT concentration at Week 12; Test type: Superiority or Other; p = 0.1515, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.75, 90% CI [0.540 to 1.044]
Statistical Analysis 4: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 4 for serum DHT concentration at Week 24; Test type: Superiority or Other; p = 0.3965, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.84, 90% CI [0.589 to 1.188]
Statistical Analysis 5: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 5 for serum Androsterone concentration at Week 12; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.42, 90% CI [0.290 to 0.615]
Statistical Analysis 6: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 6 for serum androsterone concentration at Week 24; Test type: Superiority or Other; p = 0.2494, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 1.22, 90% CI [0.916 to 1.625]
Statistical Analysis 7: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 7 for serum DHEA concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.04, 90% CI [0.023 to 0.073]
Statistical Analysis 8: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 8 for serum DHEA concentration at Week 24; Test type: Superiority or Other; p = 0.5144, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 1.24, 90% CI [0.717 to 2.137]
Statistical Analysis 9: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 9 for serum DHEA-glucuronide concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.10, 90% CI [0.055 to 0.189]
Statistical Analysis 10: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 10 for serum DHEA-glucuronide concentration at Week 24; Test type: Superiority or Other; p = 0.1329, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.55, 90% CI [0.286 to 1.060]
Statistical Analysis 11: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 11 for serum DHEA-sulfate concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.01, 90% CI [0.008 to 0.028]
Statistical Analysis 12: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 12 for serum DHEA-sulfate concentration at Week 24; Test type: Superiority or Other; p = 0.7061, ANCOVA; Adjusted mean ratio = 1.20, 90% CI [0.530 to 2.730]
Statistical Analysis 13: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 13 for serum delta-4-androstenedione concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 0.42, 90% CI [0.290 to 0.615]
Statistical Analysis 14: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 14 for serum delta-4-androstenedione concentration at Week 24; Test type: Superiority or Other; p = 0.2673, ANCOVA — [p-value comment as in outcome 4, analysis 2]; Adjusted mean ratio = 1.22, 90% CI [0.916 to 1.625]

5. Secondary Outcome: Percentage of Participants With Prostate-specific Antigen (PSA) Response
Description: The PSA response was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) criterion which is, percentage of participants with PSA less than or equal to 0.2 nanogram/milliliter at Weeks 12 and 24 after androgen deprivation.
Time Frame: Weeks 12 and 24
Population: ITT population included all the participants who were randomly assigned to the study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 30 | 28
Percentage of participants
  Week 12 | 86.7 (0.0637) | 3.6 (0.3788)
  Week 24 | 86.7 | 82.1
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for PSA response at Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Relative risk = 25.533, 90% CI [4.989 to 130.680]
Statistical Analysis 2: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 2 for PSA response at Week 24; Test type: Superiority or Other; p = 0.2319, Cochran-Mantel-Haenszel; Relative risk = 1.131, 90% CI [0.956 to 1.337]

6. Secondary Outcome: Percentage of Participants With Pathologic Complete Response (CR)
Description: Complete response is defined as a disappearance of all target lesions and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criterion.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 29 | 27
Percentage of participants | 10.3 (0.0637) | 3.7 (0.3788)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 1 for CR at Week 24; Test type: Superiority or Other; p = 0.3427, Cochran-Mantel-Haenszel; Relative risk = 2.744, 90% CI [1.018 to 5.015]

7. Secondary Outcome: Number of Participants With Tumor Expression of Androgen Receptor (AR) Regulated Genes at Week 24
Description: Tumor expression of AR regulated genes determined by real-time polymerase chain reaction (RT PCR). PCR is an in vitro method for producing large amounts of specific deoxyribonucleic acid (DNA) or ribonucleic acid fragments of defined length and sequence from small amounts of short oligonucleotide flanking sequences (primers). RT PCR is a method used for detecting the amplified DNA products from the PCR as they accumulate instead of at the end of the reaction.
Time Frame: Week 24
Population: Resullts were not reported due to insufficient data in this outcome measure.
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlation Between Molecular and Protein Expression With Intracellular Androgen Levels and Pathologic Response to Study Treatment
Description: Molecular and protein expression was correlated with intracellular androgen levels and pathologic response to study treatment.
Time Frame: Week 24
Population: Resullts were not reported due to insufficient data in this outcome measure.
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Dihydrotestosterone (DHT) Concentration in Prostate Tissue
Description: The DHT is a potent androgenic metabolite of testosterone and the concentration of DHT was measured in prostate tissues after exposure to study treatments at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picogram per milligram (pg/mg)
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Number analyzed (Participants) | 28 | 27
Picogram per milligram (pg/mg) | 4.311 (21.6213) | 2.170 (3.4589)
Statistical Analysis 1: Comparison: Abiraterone Plus Leuprolide Plus Prednisone vs Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone; Statistical Analysis 2 for DHT concentration at Week 12; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted mean ratio = 0.17, 90% CI [0.098 to 0.289]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 32
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Abiraterone Plus Leuprolide Plus Prednisone | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone
Serious Adverse Events (participants affected / at risk) | 6/30 | 7/28
Other Adverse Events (participants affected / at risk) | 30/30 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Plus Leuprolide Plus Prednisone (N=30) | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone (N=28)
Pituitary infarction (Endocrine disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hernia obstructive (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Plus Leuprolide Plus Prednisone (N=30) | Leuprolide Then Abiraterone Plus Leuprolide Plus Prednisone (N=28)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 0
Gynaecomastia (Endocrine disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Fatigue (General disorders) | 13 | 16
Irritability (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Sinusitis (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 12 | 16
Aspartate aminotransferase increased (Investigations) | 14 | 15
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Weight increased (Investigations) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 5
Libido decreased (Psychiatric disorders) | 6 | 5
Loss of libido (Psychiatric disorders) | 1 | 3
Mood altered (Psychiatric disorders) | 1 | 2
Mood swings (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 3 | 1
Pollakiuria (Renal and urinary disorders) | 5 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 1
Urine flow decreased (Renal and urinary disorders) | 3 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hot flush (Vascular disorders) | 24 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will retain the right to review all material prior to presentation or submission for publication and neither institution(s) nor Study Co-Chairs/Principal Investigator(s) is/are permitted to publish/present the results of the study, in part or in their entirety, without the written authorization of the Sponsor. The review is aimed at complying with 21CFR312.7 (non promotion of investigational drugs) as well as the intellectual property rights and commercial interests of the Sponsor.